CLINICAL TRIAL: NCT07009132
Title: Hepatic Perfusion and Liver Health as Assessed by Dual Cholate Clearance Assay in Fontan-associated Liver Disease (FALD)
Brief Title: Cholate Clearance in Fontan and Heart Failure
Status: Recruiting | Type: Observational
Sponsor: HepQuant, LLC (Industry)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: Fontan Cholate 2.0
Record Dates: First submitted 2025-05-20; First posted 2025-06-06 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Fontan; Right Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (3):
- Fontan: Patients with a Fontan diagnosis who have undergone a right heart catheterization in the past year
  Interventions: Device: Dual cholate clearance assay; Radiation: MRI
- Right Heart Failure (RHF) Controls: Non-Fontan patients with RHF (patients with normal 2-ventricle anatomy who have intermediate or elevated right-sided filling pressures (CVP) by echocardiogram)
  Interventions: Device: Dual cholate clearance assay; Radiation: MRI
- Normal Controls: Patients with normal cardiac anatomy and normal CVP (right-sided filling pressure) by echocardiogram.
  Interventions: Device: Dual cholate clearance assay; Radiation: MRI

INTERVENTIONS:
Device: Dual cholate clearance assay — Study participants are administered labeled oral and intravenous cholate, and then two blood samples are taken over 60-minutes. Serum cholate levels are measured by blood draws.
  Other Names: HepQuant dual cholate clearance assay
Radiation: MRI — Unsedated non contrast cardiac magnetic resonance imaging (MRI)

SUMMARY:
The goal of this study is to use the HepQuant dual cholate clearance assay, which has been shown to measure liver function in people with known chronic liver conditions, to assess severity of Fontan-associated liver disease (FALD).

This study aims to understand the role impaired blood flow to the liver plays in liver function in Fontan patients compared to patients with right heart failure and healthy controls. The study will also determine whether cholate clearance is a good measure to use in this population, and whether it will be able to predict clinical outcomes.

Participants will undergo a HepQuant dual cholate clearance assay and a cardiac magnetic resonance imaging (MRI) at the beginning of the study, and then data on health status will be collected for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Fontan: Adult Fontan patients ≥ 18 years of age who have undergone right heart catheterization within the past 1 year.
* RHF Controls: non-Fontan adults with two ventricle anatomy with systemic left ventricle, CVP estimate ≥ 8 mmHg and left ventricle (LV) function ≥ 50% by echocardiogram performed within the past 1 year. Can include those with congenital heart disease- repaired or unrepaired.
* Normal Controls: non-Fontan adults with normal cardiac anatomy, normal biventricular function, < moderate tricuspid regurgitation and CVP estimate < 5 mmHg by echocardiogram performed within the past 1 year.

Exclusion Criteria:

* Pregnant or breastfeeding
* Unable to comprehend and/or give informed consent
* Sensitivity to human serum albumin, or its preparations
* Participants with extensive resection of large segments of the small intestine (short gut) or severe gastroparesis
* Participants on non-selective beta blockers, angiotensin converting-enzyme (ACE) inhibitors, angiotensin receptor blockers (ARBs), ursodeoxycholic acid, cholic acid, or other bile acids who are unwilling or unable to delay taking their normal dose the morning of their dual cholate clearance testing.
* Participants on dietary supplements, bile acid sequestrants, GLP-1 agonists, narcotics, and other medications affecting gastric emptying or intestinal absorption who are unwilling or unable to delay taking or withhold as outlined in the instructions on deviating from the SHUNT test.
* Contraindication to cardiac MRI
* For RHF and normal controls: diabetes, chronic liver disease, >moderate alcohol use, BMI >30, oxygen-dependent, pulmonary hypertension22 on therapy, known porto-pulmonary hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible Fontan participants will be identified by screening the Fontan database for patients who have undergone cardiac catheterization in the past year and by searching the outpatient clinic schedule.
  Eligible RHF and normal control participants will be screened through the outpatient echo lab schedule at Hospital of the University of Pennsylvania.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Hepatic cholate clearance | Baseline
  13C-cholate and d4-cholate clearance as assessed by the dual cholate clearance test

SECONDARY OUTCOMES:
Occurrence of at Least One Heart or Liver-Related Clinical Outcome | 5 years after first cholate assay
  A patient will be considered to have a heart or liver-related clinical outcome if any of the following occur within 5 years after the first cholate assay: new-onset heart failure (defined as hospitalization for intravenous diuresis), progressive heart failure (defined as referral for heart or combined heart-liver transplant), clinically significant ascites (defined as requiring large volume paracentesis), new-onset protein-losing enteropathy, hepatocellular carcinoma, heart transplant or a combined heart and liver transplant, or death. Number of subjects with at least one of the above clinical outcomes will be captured and reported for all study groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No